CLINICAL TRIAL: NCT00196079
Title: The ASPECT Study - Asian Paclitaxel-Eluting Stent Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: April Lavender, RAC, Vice President for Regulatory Affairs, Cook
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 506
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery; stenosis; drug eluting stent; stent
MeSH Terms: conditions — Coronary Artery Disease; Constriction, Pathologic

INTERVENTIONS:
Device: Coronary stent

SUMMARY:
The ASPECT study is an Asian multicenter, randomized, controlled, triple-blinded study designed to evaluate the ability of the Cook Incorporated Paclitaxel Eluting Supra G Coronary Stent to reduce restenosis in the coronary artery.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be eligible to undergo planned treatment of a single de novo lesion in a native coronary artery.
* Patient must be an acceptable candidate for coronary artery bypass surgery.
* Patient must have given signed informed consent.
* Patient agrees to return at one month for an office visit to assess cardiovascular status and at 4-6 months for an office visit to assess cardiovascular status and for a diagnostic angiogram.

Exclusion Criteria:

* Patient is less than 18 years old.
* Patient has history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* The patient is simultaneously participating in another investigative interventional cardiovascular device or drug study.
* Patient has known hypersensitivity or contraindication to aspirin, Clopidogrel, or stainless steel, or a sensitivity to contrast dye that.
* Patient is pregnant.
* Patient has other medical condition that may cause the patient to be non-compliant with the protocol, confound the results or is associated with limited life expectancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177
Dates: Start 2000-02; Study Completion 2001-08

PRIMARY OUTCOMES:
Angiographic in-stent % diameter at follow-up.

SECONDARY OUTCOMES:
Major adverse events
Total lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Seung Jung Park, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Contact Sponsor, Bloomington, Indiana, United States